CLINICAL TRIAL: NCT05714514
Title: A Prospective, Long-term Confirmatory Follow up Trial in Highly Sensitized Patients Treated With Imlifidase or Standard of Care in the ConfIdeS (20-HMedIdeS-17) Trial
Brief Title: Survival and Dialysis Independency in Highly Sensitized Patients After Desensitization With Imlifidase and Tx of Kidneys
Acronym: ConfIdeSLTFU
Status: Active, not recruiting | Type: Observational
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-HMedIdes-25
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplantation in Highly Sensitized Patients
Keywords: Desensitization; Highly sensitized; Positive crossmatch; Unlikely to be transplanted; Renal transplantation; Deceased donor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Imlifidase administered in the ConfIdeS study
  Interventions: Drug: Imlifidase administered in the ConfIdeS study
- Best available treatment administered in the ConfIdeS study
  Interventions: Other: Best available treatment administered in the ConfIdeS study

INTERVENTIONS:
Drug: Imlifidase administered in the ConfIdeS study — Imlifidase is an immunoglobulin G (IgG)-degrading enzyme of Streptococcus pyogenes that is highly selective towards IgG. The cleavage of IgG generates one F(ab')2- and one homodimeric Fc- fragment and efficiently neutralizes Fc-mediated activities of IgG.
  Other Names: IdeS, HMED-IdeS
  Groups: Imlifidase administered in the ConfIdeS study
Other: Best available treatment administered in the ConfIdeS study — Institution-specific desensitization treatment prior to kidney transplantation in the ConfIdeS study OR remain on wait list for a more compatible organ offer if desensitization with institutional protocol is not appropriate
  Groups: Best available treatment administered in the ConfIdeS study

SUMMARY:
The goal of this follow-up study is to learn about long-term patient survival and graft function in highly sensitized patients who have received desensitization treatment with imlifidase or standard of care (SoC) in order to enable kidney transplantation in clinical study ConfIdeS (20-HMedIdeS-17, NCT04935177).

DETAILED DESCRIPTION:
This is an observational follow-up study subsequent to the ConfIdeS study (20-HMedIdeS-17, NCT04935177) in highly sensitized patients who were randomized to imlifidase or SoC desensitization prior to kidney transplantation with a deceased donor graft, or, if SoC perioperative treatment has been deemed not appropriate, wait for a more immunologically compatible organ offer.

After the patients have given written informed consent to participate in the follow-up they will be included in the study and followed until 5 years after randomization in the ConfIdeS study.

Most of the assessments in this study are already part of the follow up within SoC for these patients. During the local clinic routine follow-up visits at year 2, 3 and 5 after randomization in the ConfIdeS study, information about patient survival, wait-list status, graft survival, kidney function, and health related quality of life will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent obtained before any trial-related procedures.
2. Previous participation in the clinical trial ConfIdeS.

Exclusion Criteria:

1. Inability by the judgement of the investigator to participate in the trial for any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have participated in the clinical study ConfIdeS (20-HMedIdeS-17, NCT04935177)
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients alive and free of dialysis at 3 years | 3 years after randomization in the ConfIdeS study

SECONDARY OUTCOMES:
Proportion of patients alive and free of dialysis at 5 years | 5 years after randomization in the ConfIdeS study
Proportion of patients alive at 3 and 5 years | 3 and 5 years after randomization in the ConfIdeS study
Graft failure-free survival rates at 3 and 5 years | 3 and 5 years after randomization in the ConfIdeS study
  Graft failure-free survival is defined as time from randomization to the fist of either graft failure or death
Graft survival rates at 3 and 5 years | 3 and 5 years after randomization in the ConfIdeS study
  To be assessed in patients who were transplanted at randomization in the ConfIdeS study
Number of patients per wait-list category | 3 and 5 years after randomization in the ConfIdeS study
  The different wait-list categories are: transplanted, active, temporary inactive, inactive, or deceased
Mean estimated glomerular filtration rate (eGFR) at 3 and 5 years | 3 and 5 years after randomization in the ConfIdeS study
  eGFR is a measure of kidney function. eGFR will be calculated based on p-creatinine according to the modification of diet in renal disease (MDRD) equation. Kidney disease is characterised by a decreased eGFR value. eGFR will be set to zero, for randomized patients who do not undergo transplantation, lose their graft or die.
Proportion of patients with biopsy- and serology confirmed antibody-mediated rejection (AMR) | 3 and 5 years after randomization in the ConfIdeS study
Proportion of patients with biopsy confirmed cell-mediated rejection | 3 and 5 years after randomization in the ConfIdeS study
Treatment of graft rejection episodes | 3 and 5 years after randomization in the ConfIdeS study
  Any treatments given during rejection episodes will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Therese Åkerfeldt, Study Director — Hansa Biopharma AB
Locations (14):
- United States (14):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Northwestern University, Dept. General Surgery, Div. Transplantation, Chicago, Illinois
  - University of Chicago, Department of Surgery, Clinical Research Center, Chicago, Illinois
  - John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - New York University (NYU) Langone Transplant Institute, NYU Langone Health, New York, New York
  - Columbia University, New York, New York
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Hospital Specialty and Transplant, San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No